CLINICAL TRIAL: NCT04493762
Title: A Comparison Study of Liver Fibrosis and Its Association With Gut Microbiota in Patients With Psoriasis Vulgaris and Rheumatoid Arthritis on Methotrexate
Brief Title: Liver Fibrosis and Gut Microbiota in Patients With Psoriasis Vulgaris and Rheumatoid Arthritis on Methotrexate
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Sze-Man Wong, Associate Consultant, Queen Mary Hospital, Hong Kong
Other Study IDs: UW19-839
Record Dates: First submitted 2020-07-15; First posted 2020-07-30 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Psoriasis Vulgaris; Rheumatoid Arthritis; Fibrosis, Liver
Keywords: Methotrexate; Microbiota
MeSH Terms: conditions — Arthritis, Rheumatoid; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood (serum and plasma) and stool samples collected for this study will be saved for 3 years and stored at - 80 degree Celsius in the laboratory in Hong Kong for biomarker analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PSO/PSA: Patients diagnosed with psoriasis or psoriatic arthritis
- RA: Patients diagnosed with rheumatoid arthritis

SUMMARY:
While methotrexate (MTX) remains a treatment of choice for patients with rheumatoid arthritis (RA), psoriasis (PsO) and psoriatic arthritis (PsA), long-term MTX use has been shown to be associated with liver fibrosis and cirrhosis in these patients. In addition, gut dysbiosis has been found to be associated with liver fibrosis and cirrhosis via the gut-liver axis, underscoring the potential role of gut microbiota and bacterial translocation in the pathogenesis of chronic liver diseases in these patients.

In this study, we aim to assess the prevalence of advanced liver fibrosis or cirrhosis among these patients on MTX treatment compared to those without, using transient elastography. We also aim to identify the possible risk factor(s) for advanced liver fibrosis or cirrhosis among them. Further, we aim to characterize the difference in fecal microbiota patterns among these three groups of patients.

Using a cross-sectional, prospective cohort design, this study will enroll approximately 600 eligible patients, including 300 patients with PsO/PsA and 300 patients with RA, to examine the following hypotheses:

1. Patients on higher cumulative dose of MTX will have higher prevalence of advanced liver fibrosis or cirrhosis compared to those on lower cumulative dose of MTX;
2. Patients with MTX use will have higher prevalence of advanced liver fibrosis or cirrhosis compared to those without MTX use;
3. The fecal microbiota composition will be different between patients with and without MTX treatment; and
4. The fecal microbiota composition will be different between patients with and without advanced fibrosis/cirrhosis while on MTX treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 85 years
* Have regular follow up in Dermatology/ Rheumatology clinics of Queen Mary Hospital
* Diagnosed with PsO/PsA or RA
* Chinese ethnicity

Exclusion Criteria:

* Age below 18 years or above 85 years
* Known decompensated cirrhosis
* Pregnancy or breastfeeding
* Unstable medical illness or active infection
* Unable to provide written consent
* Unable to adhere to the protocol
* Unable to read and/or write Chinese language
* On anticoagulant/ antiplatelet treatment
* Abnormal platelet count <150
* Known disease/condition with prolonged INR/bleeding tendency

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who have regular follow up in Dermatology/ Rheumatology clinics of Queen Mary Hospital, with a diagnosis of PsO/PsA and/or RA will be identified and screened for eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-08-13 (Estimated); Primary Completion 2021-12-12 (Estimated); Study Completion 2022-12-11 (Estimated)

PRIMARY OUTCOMES:
The number of patients with advanced liver fibrosis or cirrhosis | At the time of the assessment procedure
  We will measure the number of patients with significant fibrosis (defined as having liver stiffness ≥ 7.5 kPa in transient elastography), and among those who undergo biopsy, the number of patients whose biopsy specimen is of Roenigk grades 3b or 4
The type and abundance of fecal microbiota patterns | At the time of the assessment procedure
  We will measure the type and abundance of various bacteria/viruses in specimens; alpha diversity within a specimen and beta diversity between groups of specimen; specific taxa that differ significantly between groups; and metabolic profiles and functional pathways associated with change in gut microbiota

SECONDARY OUTCOMES:
The risk factors of liver fibrosis | At the time of the assessment procedure
  Risk factors to be examined will include demographic variables such as age and gender, cumulative dose of MTX, gut dysbiosis, duration of disease, co-morbidities, hepatic steatosis, liver stiffness, and other potential factors

CONTACTS AND LOCATIONS:
Overall Officials: Sze-Man Wong, MSc, MRCP, Principal Investigator — Queen Mary Hospital, Hong Kong

IPD SHARING:
Plan to Share IPD: No